CLINICAL TRIAL: NCT02197767
Title: A Single Center Pilot Trial of Rituximab in the Treatment of Fibrillary Glomerulonephritis
Brief Title: Pilot Study of Rituximab to Treat Fibrillary Glomerulonephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Stephen B. Erickson, M.D., PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-006694
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Fibrillary Glomerulonephritis
Keywords: fibrillary glomerulonephritis; rituximab; Rituxan; MabThera; Zytux™
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Experimental): rituximab 1000 mg infusion two weeks apart for a total of two infusions. Retreated with identical rituximab 1000 mg infusion two weeks apart at six months after the first infusion for a grand total of four infusions.
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 1000 mg infusion
  Other Names: Rituxan

SUMMARY:
This pilot study is being done to see if the study medication, Rituximab, preserves kidney function after 12 months of taking the drug.

DETAILED DESCRIPTION:
This is a Phase II, open-label pilot study to determine if the use of Rituximab reduces proteinuria over a 12 month period and is there preservation of kidney function with the use of this study drug. Each patient will be treated with 2 intravenous infusions of rituximab 1000 mg, two weeks apart for a total of 2 doses. Each patient will be retreated with identical 2 intravenous infusions of rituximab, two weeks apart at 6 months after the first infusion, irrespective of cluster of differentiation (CD) 20+ cell counts. Thus, each participant will receive 4 infusions of rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Fibrillary Glomerulonephritis with diagnostic biopsy performed within the last 2 years
* Proteinuria >1 gram
* Age > 18 years but < 80 years
* Adequately controlled blood pressure (BP<140/90 mmHg in >75% of the readings) for at least 3 months prior to enrollment with the use of (angiotensin converting enzyme inhibitors (ACEi) and/or angiotensin-receptor blockers (ARB), if tolerated.
* Women must be post- menopausal, surgically sterile or practicing a medically approved method of contraception
* Able and willing to give written informed consent and comply with the requirements of the study protocol
* Adequate renal function as indicated by estimated glomerular filtration rate (GFR) > 25 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD/EPI) formula or a quantified creatinine clearance >25 mL/min, and/or serum creatinine <3.0 mg/dL in the presence of ACEi/ARB therapy
* Adequate bone marrow function, as indicated by hemoglobin >7.0 gm/dL, white count >3.0 x 10(9), platelet count >100 x 10(9)
* Negative chest x-ray within one year
* Negative serum pregnancy test (for women of child bearing age)
* Normal organ function.
* Subject agrees to use an acceptable method of birth control during treatment and for twelve months after completion of treatment
* Subject has provided written informed consent
* Subject agrees to discontinue routine use of non-steroidal anti-inflammatory drugs
* Absolute Neutrophil Count (ANC): > 1000/ mm3
* Adequate liver function, as indicated by aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and total bilirubin < 2x upper limit or normal unless related to primary disease
* Negative HBsAg and anti-hepatitis B (HBc) lab values within 1 year of signing consent

Exclusion Criteria:

* Pregnancy (determined by a serum pregnancy test for all women of childbearing potential within 7 days of treatment), or lactating.
* Inability to comply with study and/or follow-up procedures
* History of HIV (a documented positive lab value within one year of enrollment)
* Presence of active infection
* New York Heart Association Classification III or IV heart disease
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of psychiatric disorder
* At the Investigator's discretion, receipt of a live vaccine within 4 weeks prior to randomization
* At the Investigator's discretion, positive Hepatitis C serology
* Known history of diabetes mellitus or a Hemoglobin A1c result > 6.0% within 90 days prior to enrollment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B. Erickson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Erickson SB, Zand L, Nasr SH, Alexander MP, Leung N, Drosou ME, Fervenza FC. Treatment of fibrillary glomerulonephritis with rituximab: a 12-month pilot study. Nephrol Dial Transplant. 2021 Jan 1;36(1):104-110. doi: 10.1093/ndt/gfaa065. PMID 32617582

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in 24 Hour Creatinine Clearance
Description: Change in 24 hour creatinine clearance with the use of rituximab at 12 months. Creatinine clearance results are reported as milliliters/minute/patient's body surface area (mL/min/SA).
Time Frame: Day 0, Day 365
Measure: Mean (Standard Deviation); unit: mL/min/SA
Arm/Group | Rituximab
Number analyzed (Participants) | 11
mL/min/SA | 41.0 (15.52)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority; p = 0.072, t-test, 2 sided

2. Secondary Outcome: Change in Proteinuria
Description: Change in proteinuria in milligrams (mg) with the use of rituximab at 12 months.
Time Frame: Day 0, Day 365
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Rituximab
Number analyzed (Participants) | 11
mg | 2589.8 (1741.5)
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority; p = 0.068, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study until 30 days following the last administration of study treatment or study discontinuation/termination, whichever was earlier.
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT02197767/Prot_SAP_000.pdf